CLINICAL TRIAL: NCT03058627
Title: Routine Revascularization With Percutaneous Coronary Intervention in Patients With Coronary Artery Disease Undergoing Transcatheter Aortic Valve Implantation - the Nordic Aortic Valve Intervention-3 Trial
Brief Title: Revascularization in Patients Undergoing Transcatheter Aortic Valve Implantation
Acronym: NOTION-3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Engstrom (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Lund University Hospital (Other); Karolinska University Hospital (Other); Haukeland University Hospital (Other); Helsinki University Central Hospital (Other); Tampere University Hospital (Other); Oulu University Hospital (Other); Turku University Hospital (Other Government); Sahlgrenska University Hospital (Other); Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Sponsor-Investigator, Thomas Engstrom, Consultant, PhD, DMSci, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-16039929
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Aortic Valve Stenosis; TAVI; PCI
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVI only (No Intervention): TAVI is performed according to current guidelines and the choice of valve prosthesis is at the operators' discretion.
- TAVI + FFR-guided complete revascularization (Experimental): TAVI is performed according to current guidelines and the choice of transcatheter heart valve is at the operators' discretion. PCI is performed in any suitable lesion with diameter stenosis > 90% or FFR ≤ 0.80 in vessels ≥ 2.5 mm in diameter .
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — FFR guided PCI
  Arms: TAVI + FFR-guided complete revascularization

SUMMARY:
The aim of this study is to evaluate the effect of routine FFR-guided complete revascularization with PCI compared to conservative management in patients with concomitant coronary artery disease who are undergoing TAVI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Severe aortic valve stenosis and selected for TAVI by a multi-disciplinary Heart Team
3. At least one stenosis with FFR ≤ 0.80 or diameter stenosis > 90% in a coronary artery ≥ 2.5 mm in diameter

Exclusion Criteria:

1. Life expectancy < 1 year due to other severe non-cardiac disease
2. Severe renal failure with estimated glomerular filtration rate < 20 ml/min
3. No PCI-eligible coronary artery stenosis, but rotablation is allowed
4. Admitted with a new acute coronary syndrome (ST-elevation myocardial infarction (STEMI) or non-STEMI) within 14 days
5. Significant stenosis in left main stenosis or ostial left anterior descending artery (LAD) + ostial left circumflex artery (LCx))
6. Only stenoses with thrombolysis in myocardial infarction grad < 3
7. Potential pregnancy
8. Known allergy towards P2Y12 receptor antagonists, heparin or contrast medium
9. More than one chronic total occlusion (CTO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality, myocardial infarction, or urgent revascularization | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing all-cause mortality, myocardial infarction, or urgent PCI

SECONDARY OUTCOMES:
All cause mortality | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing all cause mortality
Myocardial infarction | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing myocardial infarction
Urgent revascularization | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing urgent revascularization
All cause mortality or myocardial infarction | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing all cause mortality or myocardial infarction
Cardiovascular mortality | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing cardiovascular mortality
Cardiovascular mortality, myocardial infarction, or urgent PCI | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing cardiovascular mortality, myocardial infarction, or urgent PCI
Cardiovascular mortality or myocardial infarction | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing cardiovascular mortality or myocardial infarction
Admission for new onset of heart failure | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing admission for new onset of heart failure
Peri-procedural (PCI) myocardial infarction | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing peri-procedural (PCI) myocardial infarction
Peri-procedural (TAVI) myocardial infarction | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing peri-procedural (TAVI) myocardial infarction
Any revascularization | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing any revascularization
Stroke or transient ischemic attack (TIA) | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing stroke or transient ischemic attack (TIA)
Angina status (Seattle questionnaire), CCS and NYHA class | 30 days and 1 year
  Number of patients experiencing CCS and NYHA class
Bleeding | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing bleeding
Quality of Life | 30 days and 1 year
  Number of patients experiencing improvement in Quality of life
Acute kidney injury | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing acute kidney injury
Target vessel revascularization | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing target vessel revascularization
Target lession revascularization | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing target lession revascularization
Cost effectiveness analysis | Until the last included patients have been followed for 1 year after the TAVI
  Cost effectiveness analysis
Stent thrombosis | Until the last included patients have been followed for 1 year after the TAVI
  Number of patients experiencing stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrøm, MD, DMSC, PhD, Study Chair — Rigshospitalet University Hospital, Denmark; Jacob Lønborg, MD, DMSC, PhD, Principal Investigator — Rigshospitalet University Hospital, Denmark; Lars Søndergaard, MD, DMSc, PhD, Study Chair — Rigshospitalet University Hospital, Denmark
Locations (12):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Department of Cardiology, Skejby University Hospital, Aarhus
  - Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - Department of Cardiology, Odense University Hospital, Odense
- Finland (4):
  - Helsinki University Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Riga University Hospital, Riga, Latvia
- Sweden (3):
  - Sahlgrenska, Gothenburg
  - Lund University Hospital, Lund
  - Karolinska, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jorgensen TH, Engstrom T, Jabbari R, Glinge C, Sabbah M, Veien KT, Niemela M, Freeman P, Linder R, Sorensen R, Holmvang L, Ioanes D, Terkelsen CJ, Ellert-Gregersen J, Christiansen E, Eftekhari A, Piuhola J, Kajander O, Koul S, Savontaus M, Karjalainen P, Sondergaard L, De Backer O, Lonborg J. Fractional Flow Reserve to Guide Revascularization in Patients With Coronary Artery Disease Undergoing TAVR. JACC Cardiovasc Interv. 2025 Dec 8;18(23):2925-2936. doi: 10.1016/j.jcin.2025.10.015. PMID 41371788
- [Derived] Lonborg J, Jabbari R, Sabbah M, Veien KT, Niemela M, Freeman P, Linder R, Ioanes D, Terkelsen CJ, Kajander OA, Koul S, Savontaus M, Karjalainen P, Erglis A, Minkkinen M, Sorensen R, Tilsted HH, Holmvang L, Bieliauskas G, Ellert J, Piuhola J, Eftekhari A, Angeras O, Ruck A, Christiansen EH, Jorgensen T, Ozbek BT, Glinge C, Sondergaard L, De Backer O, Engstrom T; NOTION-3 Study Group. PCI in Patients Undergoing Transcatheter Aortic-Valve Implantation. N Engl J Med. 2024 Dec 12;391(23):2189-2200. doi: 10.1056/NEJMoa2401513. Epub 2024 Aug 31. PMID 39216095